CLINICAL TRIAL: NCT00024258
Title: Phase II Study of Arsenic Trioxide in Neuroblastoma and Other Pediatric Solid Tumors
Brief Title: Arsenic Trioxide in Treating Patients With Advanced Neuroblastoma or Other Childhood Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-042; P30CA008748 (NIH); MSKCC-01042; CTI-1059; NCI-G01-2014
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-10

CONDITIONS: Brain and Central Nervous System Tumors; Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Kidney Cancer; Liver Cancer; Neuroblastoma; Ovarian Cancer; Retinoblastoma; Sarcoma
Keywords: metastatic osteosarcoma; recurrent childhood rhabdomyosarcoma; regional neuroblastoma; disseminated neuroblastoma; stage 4S neuroblastoma; recurrent neuroblastoma; stage III childhood liver cancer; stage IV childhood liver cancer; recurrent childhood liver cancer; childhood hepatoblastoma; stage III Wilms tumor; stage IV Wilms tumor; stage V Wilms tumor; recurrent Wilms tumor and other childhood kidney tumors; intraocular retinoblastoma; extraocular retinoblastoma; recurrent retinoblastoma; recurrent osteosarcoma; childhood germ cell tumor; metastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; localized unresectable neuroblastoma; previously untreated childhood rhabdomyosarcoma; childhood desmoplastic small round cell tumor; untreated childhood medulloblastoma; recurrent childhood medulloblastoma; previously treated childhood rhabdomyosarcoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; childhood teratoma; childhood malignant testicular germ cell tumor; childhood malignant ovarian germ cell tumor; childhood extragonadal germ cell tumor; recurrent childhood malignant germ cell tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Kidney Neoplasms; Liver Neoplasms; Neuroblastoma; Ovarian Neoplasms; Retinoblastoma; Sarcoma; Osteosarcoma; Hepatoblastoma; Wilms Tumor; Desmoplastic Small Round Cell Tumor; Medulloblastoma; Neuroectodermal Tumors, Primitive, Peripheral; Teratoma; Testicular Neoplasms; Ovarian Germ Cell Cancer | interventions — Arsenic Trioxide

ARMS (1):
- Arsenic Trioxide (Experimental): Patients receive arsenic trioxide IV over 1-4 hours on days 1-5 and 8-12. Treatment repeats every 28 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 2-3 months for 1 year and then annually thereafter.
  Interventions: Drug: arsenic trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of arsenic trioxide in treating children who have advanced neuroblastoma or other solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rates of patients with advanced neuroblastoma or other pediatric solid tumors treated with arsenic trioxide.
* Determine the toxicity of this drug in these patients.

OUTLINE: Patients are stratified according to type of disease (neuroblastoma with progressive disease vs neuroblastoma with stable refractory disease vs other solid tumor).

Patients receive arsenic trioxide IV over 1-4 hours on days 1-5 and 8-12. Treatment repeats every 28 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2-3 months for 1 year and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed neuroblastoma or other pediatric solid tumor (nonmyeloid and nonlymphoid) including the following:

  * Ewing's family of tumors/primitive neuroectodermal tumor
  * Retinoblastoma
  * Nephroblastoma
  * Osteosarcoma
  * Rhabdomyosarcoma
  * Desmoplastic small round-cell tumor
  * Hepatoblastoma
  * Germ cell tumors
  * Medulloblastoma
* Relapsed from or resistant to prior standard anticancer therapy and/or no known standard therapy available
* Measurable disease (e.g., solid mass with definable dimensions) OR
* Evaluable disease (e.g., bone marrow involvement or malignant pleural effusion)

PATIENT CHARACTERISTICS:

Age:

* 40 and under

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2.5 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 2.5 times ULN

Cardiovascular:

* Absolute QT interval no greater than 460 msec in the presence of adequate potassium and magnesium levels

Other:

* No pre-existing neurotoxicity/neuropathy grade 2 or greater
* No pre-existing convulsive disorder
* No active serious infections uncontrolled by antibiotics
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* More than 3 weeks since prior cytotoxic chemotherapy
* No other concurrent cytotoxic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Concurrent radiotherapy allowed provided measurable or evaluable disease exists outside radiation field

Surgery:

* Not specified

Other:

* No other concurrent investigational agents

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2001-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian H. Kushner, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arsenic Trioxide
Started | 22
Completed | 13
Not Completed | 9
Not completed — Withdrawal by Subject | 1
Not completed — Disease Progression | 8

BASELINE CHARACTERISTICS:
Arm/Group | Arsenic Trioxide
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Response Rate After Every 3 Courses During Treatment and Then Every 2-3 Months for 1 Year After Completion of Treatment
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Arsenic Trioxide
Number analyzed (Participants) | 21
participants
  Progression of Disease | 16
  Stable Disease | 5

ADVERSE EVENTS:
Arm/Group | Arsenic Trioxide
Serious Adverse Events (participants affected / at risk) | 12/22
Other Adverse Events (participants affected / at risk) | 14/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arsenic Trioxide (N=22)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Infection NOS (Infections and infestations) | 4 (4)
Neuralgia (Nervous system disorders) | 1 (1)
Neutrophil count decrease (Investigations) | 3 (4)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arsenic Trioxide (N=22)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (15)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dry Eye (Eye disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema (General disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Gastrointestinal other (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Infection w/o neutropenia (Infections and infestations) | 4 (4)
White blood cell decreased (Investigations) | 1 (4)
Anxiety (Psychiatric disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Neurology, other (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (6)
Pain, other (General disorders) | 3 (4)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes